CLINICAL TRIAL: NCT03182777
Title: Safety of Local Dental Anesthesia in Patients With Cardiac Channelopathies
Acronym: SLDAPCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Itamara Lucia Itagiba Neves, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Odonto-Canalopatias
Record Dates: First submitted 2015-10-15; First posted 2017-06-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Channelopathies; Brugada Syndrome; Long QT Syndrome; Ventricular, Tachycardia
Keywords: arrhythmias, cardiac; channelopathies; death, sudden; genetic testing; electrocardiography, ambulatory; anesthesia, local; dentistry
MeSH Terms: conditions — Channelopathies; Brugada Syndrome; Long QT Syndrome; Tachycardia, Ventricular; Arrhythmias, Cardiac; Death, Sudden

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine with epinephrine (Active Comparator): Application of local dental anesthesia with two cartridges (3,6 mL) of lidocaine 2% with epinephrine 1:100.000 for dental restorative procedures in patients with cardiac channelopathies.
  Interventions: Procedure: Dental restorative procedure
- Lidocaine (Active Comparator): Application of local dental anesthesia with two cartridges (3,6 mL) of lidocaine 2% without vasoconstrictor for dental restorative procedures in patients with cardiac channelopathies.
  Interventions: Procedure: Dental restorative procedure

INTERVENTIONS:
Procedure: Dental restorative procedure — Infiltration of two cartridges (3.6 mL) of local anesthetics with 2% lidocaine with or without epinephrine 1:100,000, in two sessions with an interval of seven days between them, in oral mucosa in patients with cardiac channelopathies.

SUMMARY:
Patients with cardiac channelopathies needing restorative dental treatment will be included in two sessions of the study, using local dental anesthetic: lidocaine 2% with epinephrine and lidocaine 2% without vasoconstrictor. The safety of the use of two cartridges (3.6 mL) will be evaluated. The patients will be their own control and will be assessed by Holter monitoring for 28 hours, blood pressure measurement and anxiety measuring.

DETAILED DESCRIPTION:
Patients of Heart Institute of the University of São Paulo with inherited cardiac channelopathies will be included, considering the criteria for inclusion and non-inclusion, after reading and signing the informed consent.

They will undergo dental restorative treatment in two sessions, in the morning period, with an interval of at least seven days (wash-out) between them, and the patients will be their own control.

In the first session, after randomization, patients will receive lidocaine 2% without vasoconstrictor (LSA) or lidocaine 2% with 1: 100,000 epinephrine (LCA) (cross-over), resulting in two conditions: with adrenaline and without adrenaline.

The randomization of the anesthetic solution will be performed by the main researcher, being blind to the performer researcher and to the patient.

The injected volume will be 3.6 mL (2 cartridges) of the anesthetic solution, using blocking technique of the inferior alveolar nerve.

The patients will be monitored by Holter for 28 hours starting one hour before the procedure, for registration and analysis of cardiac electrical activity during the two sessions. Blood pressure will be monitored with digital sphygmomanometer and anxiety will be measured with Facial Image Scale, both on three occasions: at the beginning of the baseline periods, before starting application of anesthesia and at the end of the proceedings. The results will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any channelopathies below, kept on optimal drug therapy, with or without ICD:

Brugada Syndrome, Long QT Syndrome and Catecholaminergic Polymorphic Ventricular Tachycardia

* Dental caries or unsatisfactory restorations in the mandible, indicating restorative dental treatment

Exclusion Criteria:

* Patients allergic to lidocaine
* Patients undergoing ICD therapy for less than three months
* Patients with recurrent syncope in the last three months
* Patients with sustained arrhythmias documented for less than 3 months
* Have received epinephrine in the last 24 hours

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-05; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
No sustained ventricular tachycardia | during dental procedures
  No life-threatening arrhythmias and clinical signs and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Itamara LI Neves, PhD, Principal Investigator — Instituto do Coração do HCFMUSP; Ana CG Oliveira, S, Study Chair — Instituto do Coração do HCFMUSP; Ricardo S Neves, PhD, Study Director — Instituto do Coração do HCFMUSP; Luciana Sacilotto, S, Study Chair — Instituto do Coração do HCFMUSP; Francisco CC Darrieux, PhD, Study Chair — Instituto do Coração do HCFMUSP; Maurício I Scanavacca, PhD, Study Director — Instituto do Coração do HCFMUSP; Denise Hachul, PhD, Study Chair — Instituto do Coração do HCFMUSP; Cesar J Gruppi, PhD, Study Director — Instituto do Coração do HCFMUSP
Locations (1):
- Heart Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
After thesis defense, the IPD will be available on the Portal Digital Library of Theses and Dissertations of the University of São Paulo (http://www.teses.usp.br/index.php?option=com_jumi&fileid=12&Itemid=77&lang=pt-br), in a PDF file.

REFERENCES:
- [Background] Amin AS, Asghari-Roodsari A, Tan HL. Cardiac sodium channelopathies. Pflugers Arch. 2010 Jul;460(2):223-37. doi: 10.1007/s00424-009-0761-0. Epub 2009 Nov 29. PMID 20091048
- [Background] Kauferstein S, Kiehne N, Neumann T, Pitschner HF, Bratzke H. Cardiac gene defects can cause sudden cardiac death in young people. Dtsch Arztebl Int. 2009 Jan;106(4):41-7. doi: 10.3238/arztebl.2009.0041. Epub 2009 Jan 23. PMID 19564966
- [Background] Perusse R, Goulet JP, Turcotte JY. Contraindications to vasoconstrictors in dentistry: Part I. Cardiovascular diseases. Oral Surg Oral Med Oral Pathol. 1992 Nov;74(5):679-86. doi: 10.1016/0030-4220(92)90365-w. PMID 1437073
- [Background] Groban L, Deal DD, Vernon JC, James RL, Butterworth J. Ventricular arrhythmias with or without programmed electrical stimulation after incremental overdosage with lidocaine, bupivacaine, levobupivacaine, and ropivacaine. Anesth Analg. 2000 Nov;91(5):1103-11. doi: 10.1097/00000539-200011000-00011. PMID 11049891
- [Background] Jowett NI, Cabot LB. Patients with cardiac disease: considerations for the dental practitioner. Br Dent J. 2000 Sep 23;189(6):297-302. doi: 10.1038/sj.bdj.4800750. PMID 11060950
- [Background] Rochford C, Seldin RD. Review and management of the dental patient with Long QT syndrome (LQTS). Anesth Prog. 2009 Summer;56(2):42-8. doi: 10.2344/0003-3006-56.2.42. PMID 19642718
- [Background] Buchanan H, Niven N. Validation of a Facial Image Scale to assess child dental anxiety. Int J Paediatr Dent. 2002 Jan;12(1):47-52. PMID 11853248
- [Background] Naftalin LW, Yagiela JA. Vasoconstrictors: indications and precautions. Dent Clin North Am. 2002 Oct;46(4):733-46, ix. doi: 10.1016/s0011-8532(02)00021-6. PMID 12436828
- [Background] Pallasch TJ. Vasoconstrictors and the heart. J Calif Dent Assoc. 1998 Sep;26(9):668-73, 676. PMID 9879236
- [Background] Finder RL, Moore PA. Adverse drug reactions to local anesthesia. Dent Clin North Am. 2002 Oct;46(4):747-57, x. doi: 10.1016/s0011-8532(02)00018-6. PMID 12436829
- [Background] Goulet JP, Perusse R, Turcotte JY. Contraindications to vasoconstrictors in dentistry: Part III. Pharmacologic interactions. Oral Surg Oral Med Oral Pathol. 1992 Nov;74(5):692-7. doi: 10.1016/0030-4220(92)90367-y. PMID 1359489
- [Background] Brown RS, Rhodus NL. Epinephrine and local anesthesia revisited. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Oct;100(4):401-8. doi: 10.1016/j.tripleo.2005.05.074. No abstract available. PMID 16182160
- [Background] Hersh EV, Giannakopoulos H. Beta-adrenergic blocking agents and dental vasoconstrictors. Dent Clin North Am. 2010 Oct;54(4):687-96. doi: 10.1016/j.cden.2010.06.009. PMID 20831932
- [Background] Neves RS, Neves IL, Giorgi DM, Grupi CJ, Cesar LA, Hueb W, Grinberg M. Effects of epinephrine in local dental anesthesia in patients with coronary artery disease. Arq Bras Cardiol. 2007 May;88(5):545-51. doi: 10.1590/s0066-782x2007000500008. English, Portuguese. PMID 17589629
- [Background] Yagiela JA. Adverse drug interactions in dental practice: interactions associated with vasoconstrictors. Part V of a series. J Am Dent Assoc. 1999 May;130(5):701-9. doi: 10.14219/jada.archive.1999.0280. PMID 10332135
- [Background] Caceres MT, Ludovice AC, Brito FS, Darrieux FC, Neves RS, Scanavacca MI, Sosa EA, Hachul DT. Effect of local anesthetics with and without vasoconstrictor agent in patients with ventricular arrhythmias. Arq Bras Cardiol. 2008 Sep;91(3):128-33, 142-7. doi: 10.1590/s0066-782x2008001500002. English, Portuguese. PMID 18853053
- [Background] Theodotou N, Cillo JE Jr. Brugada syndrome (sudden unexpected death syndrome): perioperative and anesthetic management in oral and maxillofacial surgery. J Oral Maxillofac Surg. 2009 Sep;67(9):2021-5. doi: 10.1016/j.joms.2009.04.043. No abstract available. PMID 19686944
- [Background] Ackerman MJ, Khositseth A, Tester DJ, Hejlik JB, Shen WK, Porter CB. Epinephrine-induced QT interval prolongation: a gene-specific paradoxical response in congenital long QT syndrome. Mayo Clin Proc. 2002 May;77(5):413-21. doi: 10.4065/77.5.413. PMID 12004990
- [Background] Wynn RL. Articaine 4% with 1:200,000 epinephrine: an acceptable option for patients with long QT syndrome. Gen Dent. 2007 May-Jun;55(3):176-8. No abstract available. PMID 17511356
- [Background] Middlehurst RJ, Gibbs A, Walton G. Cardiovascular risk: the safety of local anesthesia, vasoconstrictors, and sedation in heart disease. Anesth Prog. 1999 Fall;46(4):118-23. PMID 11692352
- [Background] Fujiki A, Nishida K, Mizumaki K, Nagasawa H, Shimono M, Inoue H. Spontaneous onset of torsade de pointes in long-QT syndrome and the role of sympathovagal imbalance. Jpn Circ J. 2001 Dec;65(12):1087-90. doi: 10.1253/jcj.65.1087. PMID 11768004
- [Background] Monteforte N, Napolitano C, Priori SG. Genetics and arrhythmias: diagnostic and prognostic applications. Rev Esp Cardiol (Engl Ed). 2012 Mar;65(3):278-86. doi: 10.1016/j.recesp.2011.10.008. Epub 2012 Jan 14. English, Spanish. PMID 22245453
- [Background] Ernesto C, Cruz FE, Lima FS, Coutinho JL, Silva R, Urmenyi TP, Carvalho AC, Rondinelli E. Investigation of ion channel gene variants in patients with long QT syndrome. Arq Bras Cardiol. 2011 Mar;96(3):172-8. doi: 10.1590/s0066-782x2011005000015. Epub 2011 Feb 4. English, Portuguese, Spanish. PMID 21308345
- [Background] Meyer JS, Mehdirad A, Salem BI, Kulikowska A, Kulikowski P. Sudden arrhythmia death syndrome: importance of the long QT syndrome. Am Fam Physician. 2003 Aug 1;68(3):483-8. PMID 12924831
- [Derived] Oliveira ACG, Neves ILI, Sacilotto L, Olivetti NQS, Santos-Paul MAD, Montano TCP, Carvalho CMA, Wu TC, Grupi CJ, Barbosa SA, Pastore CA, Samesima N, Hachul DT, Scanavacca MI, Neves RS, Darrieux FCC. Is It Safe for Patients With Cardiac Channelopathies to Undergo Routine Dental Care? Experience From a Single-Center Study. J Am Heart Assoc. 2019 Aug 6;8(15):e012361. doi: 10.1161/JAHA.119.012361. Epub 2019 Jul 19. PMID 31319747